CLINICAL TRIAL: NCT06115746
Title: A Randomized Clinical Trial of a Novel Drug Education and Diversion Program (iDECIDE) for Middle and High School Students
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Massachusetts Department of Health (Other Government)
Responsible Party: Principal Investigator, Randi Melissa Schuster, Associate Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2023P000808; INTF2400H78500224455 (Other Grant/Funding Number: Massachusetts Department of Public Health)
Record Dates: First submitted 2023-10-30; First posted 2023-11-03 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Substance Use; Harm Reduction; Adolescent Behavior
Keywords: Adolescent; Diversion program; iDECIDE; Tier 2; School; Substance use prevention; Addiction; Early intervention; Targeted prevention
MeSH Terms: conditions — Substance-Related Disorders; Harm Reduction; Adolescent Behavior; Behavior, Addictive

STUDY DESIGN:
Intervention Model Description: Approximately 300 participants will be enrolled into a two-arm, assessor-blind, randomized controlled trial to compare substance use outcomes (i.e., knowledge, behavior, and attitudes) across a one-year follow-up period in adolescents randomly assigned to the iDECIDE drug curriculum or the waitlist control group.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Eligible participants will be randomly assigned at the end of the baseline visit in a 1:1 ratio, in blocks of 6, to either a waitlist control group or the iDECIDE curriculum group. Randomization will be stratified by substance use frequency. Treatment will be assigned according to study number, assigned sequentially to eligible participants who enroll in the trial and attend the baseline visit. Investigators and outcome assessors will be fully blinded to allocation across the two arms. Facilitators of the iDECIDE curriculum will not be involved with the data outcome assessments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- iDECIDE (Experimental): Participants will…
  1. Receive 4 weekly sessions of the iDECIDE drug curriculum.
  2. Complete assessments and questionnaires, including self-reports of substance use and 4 urinalysis visits.
  3. Be video recorded for quality control.
  Interventions: Behavioral: iDECIDE
- Waitlist Control Group (No Intervention): Participants will…
  1. Not receive the iDECIDE curriculum during the weekly visits. They can choose to self-enroll in the iDECIDE curriculum at their one-month follow up visit.
  2. Undergo symptom monitoring during the weekly visits.
  3. Complete assessments and questionnaires, including self-reports of substance use and 4 urinalysis visits.

INTERVENTIONS:
Behavioral: iDECIDE — iDECIDE is a 4-session drug education and diversion program that addresses topics such as the neurobiology and addiction, adolescent brain development, industry tactics, motives for using substances, risk and protective factors, identifying triggers, healthy alternatives, core values, and long-term goal setting. These topics are taught via facilitated discussions, videos, worksheets, and handouts. The iDECIDE drug curriculum will be delivered weekly for 4 weeks via videoconference or in-person visits. Each session typically takes 60-75 minutes. For this study, facilitators are members of study staff.
  Other Names: Drug Education Curriculum: Intervention, Diversion, and Empowerment
  Arms: iDECIDE

SUMMARY:
The primary goal of this study is to test the effectiveness of the iDECIDE (Drug Education Curriculum: Intervention, Diversion, and Empowerment) curriculum, a novel drug education and diversion program, in approximately 300 middle and high school students, who have violated their school substance use policies in the past month, as an alternative to punitive school responses for school-based substance use infractions. This randomized controlled trial will test the hypothesis that adolescents randomized to the iDECIDE curriculum will have improved substance use outcomes (i.e., knowledge, attitudes, and behavior) compared to adolescents in a waitlist control group. The outcomes of this study will measure knowledge of drug effects and brain development, perceptions of harm from substance use, willingness to quit or reduce use, and substance use behavior.

DETAILED DESCRIPTION:
This study will be a two-arm, assessor-blind, randomized controlled trial enrolling approximately 300 middle and high school students who have recently violated a school substance use policy. Participants will be followed over a one-year period. Participants will be randomly assigned to either four-weeks of iDECIDE or a waitlist control group. Participants assigned to receive iDECIDE will receive a drug education curriculum developed to provide behavioral support and psychoeducation via videoconference or in-person visits. The purpose of iDECIDE is to provide students with the knowledge and skills they need to make healthy decisions regarding substance use. Participants in the waitlist control group will undergo symptom and substance use monitoring only, until completion of the one-month follow-up visit at which point they will be offered the opportunity to enroll in the iDECIDE curriculum, if desired. Data collection will occur during nine visits over the span of approximately one year, including one randomization baseline visit, four weekly visits during the intervention phase of the study during which time participants will participate in either iDECIDE or monitoring, and then four follow-up visits. The follow-up visits will occur at approximately one week, one month, six months, and one year following the end-of-intervention. Participants in both arms will complete questionnaires and assessments conducted by raters blinded to study arm assignment. Primary outcomes (knowledge of drug effects, knowledge of brain development and neurobiology of addiction, readiness to quit, perceptions of harm, and frequency of substance use) will be assessed at visit 1 (baseline), visit 5 (end-of-intervention), visit 6 (one week follow-up), and visit 7 (one month follow-up). Participants will be compensated for session attendance and provision of urine samples.

ELIGIBILITY:
Inclusion Criteria:

1. Currently enrolled in middle or high school;
2. Violated school substance use policy within approximately the past month at the time of screening;
3. Have a parent or legal guardian who is able and willing to provide written informed consent (if under the age of 18);
4. Competent and willing to provide written informed assent (if under the age of 18) or written informed consent (if age 18 or older);
5. Able to commit to 9 study visits over approximately one year;
6. Able to safely participate in the protocol and appropriate for outpatient level of care, in the opinion of the investigator;
7. Has access to a reliable internet connection and a device that can run Zoom;
8. Able to read and write comfortably in one of the languages spoken by study staff.

Exclusion Criteria:

1. Ever received substance use treatment in an inpatient or specialty care setting;
2. Ever engaged in intravenous (IV) drug use;
3. Current daily use of alcohol, non-medical benzodiazepines, and/or opioid use.

Ages: 9 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-11-17 (Actual); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Knowledge of Drug Effects and Brain Development | Baseline to 1-month follow-up (primary), 6-month and 1-year follow-up (exploratory)
  Knowledge of drug effects and brain development will be measured with a multiple choice questionnaire that assesses knowledge taught in the iDECIDE curriculum, including neurobiology of addiction, side effects of substance, and industry tactics to market substances to young audiences.
Frequency of Substance Use | Baseline to 1-month follow-up (primary), 6-month and 1-year follow-up (exploratory)
  The Timeline Follow-Back (TLFB) will be used to measure number of days the participant used a substance, which substances were used, and the frequency of which substances were used. The initial TLFB at the baseline visit will measure substances used in the past 90 days, while the interim TLFB will measure substances used since each subsequent visit. Participants will also provide a urine sample at study visits 1, 5, 6, 7 to qualitatively screen for substances including amphetamines, cocaine, barbiturates, methamphetamines, benzodiazepines, opiates, marijuana, phencyclidine, propoxyphene, and methaqualone using a urine 10-panel. There will also be an assay to quantitate levels of cotinine and creatinine-adjusted carboxy THC at baseline, end-of-intervention, one-week follow-up, and one-month follow-up. The primary outcome will be change in frequency of past week use (number of days) for the substance used most frequently at baseline.
Readiness to Quit or Reduce Substance Use | Baseline to 1-month follow-up (primary), 6-month and 1-year follow-up (exploratory)
  Participants will complete a Readiness Ruler to determine how ready they are to reduce their substance use on a scale from 1 (not at all ready) to 10 (very ready).
Perceived Harm of Substance Use | Baseline to 1-month follow-up (primary), 6-month and 1-year follow-up (exploratory)
  The Perceived Harm of Substance Use measure was modified from the 2010 National Survey on Drug Use and Health. Participants will assess their perceived harm of various forms of substance use using four response categories that range from no risk to great risk.

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie reported results (after de-identification [text, tables, figures, and appendices]), and the study protocol, statistical analysis plan, analytic code, and informed consent form will be made available to researchers who provide a methodologically sound proposal beginning 3 months and ending 5 years following article publication to achieve aims in the approved proposal. Proposals should be directed to rschuster@harvard.mgh.edu. To gain access, data requestors will need to sign a data access agreement.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Beginning 3 months and ending 5 years following article publication
Access Criteria: Researchers who provide a methodologically sound proposal to achieve aims in the approved proposal. Data access agreement required.

REFERENCES:
- [Background] Liu J, Butler R, Turncliff A, Gray C, Lynch S, Whittaker J, Iroegbulem V, Howell D, Schuster RM. An Urgent Need for School-Based Diversion Programs for Adolescent Substance Use: A Statewide Survey of School Personnel. J Adolesc Health. 2023 Sep;73(3):428-436. doi: 10.1016/j.jadohealth.2023.04.006. Epub 2023 Jun 15. PMID 37318411
- [Background] Schuster RM, Cather C, Pachas GN, Nielsen L, Iroegbulem V, Dufour J, Potter K, Levy S, Gray KM, Evins AE. A randomized controlled trial of varenicline and brief behavioral counseling delivered by lay counselors for adolescent vaping cessation: Study protocol. Front Psychiatry. 2023 Mar 15;14:1083791. doi: 10.3389/fpsyt.2023.1083791. eCollection 2023. PMID 37009114